CLINICAL TRIAL: NCT02373150
Title: A Phase 1, Randomised, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Study to Assess the Safety, Tolerability and Pharmacokinetics of Imeglimin in Healthy Japanese Subjects
Brief Title: Safety, Tolerability and PK of Imeglimin in Japanese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Poxel SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PXL008-011
Record Dates: First submitted 2015-02-02; First posted 2015-02-26 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — imeglimin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A1 (Experimental): Dose 1 or placebo
  Interventions: Drug: Imeglimin; Drug: Placebo
- Group A2 (Experimental): Dose 2 or placebo
  Interventions: Drug: Imeglimin; Drug: Placebo
- Group A3 (Experimental): Dose 3 or placebo
  Interventions: Drug: Imeglimin; Drug: Placebo

INTERVENTIONS:
Drug: Imeglimin
Drug: Placebo

SUMMARY:
This study will assess the pharmacokinetics of single and repeated doses of imeglimin in healthy Japanese subjects, and the safety and tolerability of single and repeated doses of imeglimin in healthy Japanese subjects.

DETAILED DESCRIPTION:
Combined single and repeated dose groups with 3 escalating doses

ELIGIBILITY:
Inclusion Criteria:

* Male or female Japanese subjects, deemed healthy on the basis of a clinical history, physical examination, ECG, vital signs, and laboratory tests of blood and urine
* Body mass index in the range 18.0-25.0 kg/m2
* Willing to use reliable contraception
* Able to give fully informed written consent.

Exclusion Criteria:

* Pregnant or lactating woman, or sexually active woman of child-bearing potential not using reliable contraception
* Clinically relevant abnormal findings at the screening assessment
* Clinically significant vital signs outside the acceptable range at screening
* Clinically relevant abnormal medical history, surgery or concurrent medical condition
* Acute or chronic illness
* Estimated glomerular filtration rate less than 80 mL/min/1.73 m2
* Severe adverse reaction to any drug or sensitivity to the trial medication or its components
* Significant food allergy; vegetarian or vegan
* Use of vitamins, herbal medicines, or over-the-counter medication (with the exception of paracetamol [acetaminophen]) within 7 days before first dose of trial medication, or prescribed medication during the 14 days before first dose of trial medication
* Participation in other clinical trials of unlicensed or prescription medicines, or loss of more than 400 mL blood, within the 3 months before first dose of trial medication
* Drug or alcohol abuse
* Smoking of more than 5 cigarettes daily
* Possibility that subject will not cooperate
* Positive test for hepatitis B & C, HIV
* Objection by a General Practitioner.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2015-02; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
PK parameters of imeglimin after single and repeated doses: - Cmax: peak plasma concentration after dosing, AUC0-∞: area under the concentration-time curve from 0 extrapolated to infinite time, - Tmax: time of peak plasma concentration of imeglimin | From baseline to Day 13
  * Cmax: peak plasma concentration after dosing
  * AUC0-∞: area under the concentration-time curve from 0 extrapolated to infinite time
  * AUC0-t: area under the concentration-time curve from 0 to the time of last quantifiable concentration
  * Tmax: time of peak plasma concentration of imeglimin
Safety and tolerability of imeglimin: laboratory assessments | From baseline to Day 13
  * routine hematology, biochemistry, coagulation and urinalysis
  * physical examination
  * 12-lead ECG
  * vital signs
  * capillary glucose
  * incidence of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Hammersmith Medicines Research (HMR), London, United Kingdom